CLINICAL TRIAL: NCT00154284
Title: A 12 Month, Multicenter, Randomized, Parallel, Open-label Study, to Evaluate Renal Function and Efficacy of Everolimus With Basiliximab and Cyclosporine Microemulsion Discontinuation at 3 Month Post-transplant Versus Minimization, in de Novo Kidney Transplant Recipients
Brief Title: Everolimus in a Cyclosporine Microemulsion-free Regimen Compared to a Low-dose Cyclosporine Microemulsion Regimen, in de Novo Kidney Transplant Patients
Acronym: CERTES02
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: novartis, novartis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001A2419; CRAD001A2423 (Other: Novartis Pharmaceuticals); NCT00170807 (obsolete NCT alias)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2011-03-11 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-07

CONDITIONS: Organ Transplantation, Renal Transplantation
Keywords: Renal transplantation,; everolimus,; immunosuppressants,; basiliximab,; cyclosporine microemulsion discontinuation, cyclosporine microemulsion minimization
MeSH Terms: interventions — Everolimus; Cyclosporine; Steroids; Prednisone; Basiliximab

ARMS (2):
- Everolimus (Certican) with Cyclosporine (Neoral) Continuation (Active Comparator): Patients were treated with everolimus and cyclosporine for 3 months post-transplantation. Everolimus (Certican) was administered orally, in two divided doses (b.i.d), and at the same time as Cyclosporine (Neoral). Everolimus (Certican) dose was adjusted in order to maintain a trough level between 3 and 8 ng/mL until randomization. After randomization the target trough range remained at 3 - 8 ng/mL in the cyclosporine (Neoral) continuation groups for a period of 9 months. Each patient was administered i.v. prednisone (or equivalent) pre- or intra-operatively according to center practice.
  Interventions: Drug: Everolimus (Certican); Drug: Cyclosporine (Neoral); Drug: Steroid; Drug: Basiliximab (Simulect)
- Everolimus (Certican) with Cyclosporine (Neoral) Withdrawal (Experimental): Patients were treated with everolimus and cyclosporine for 3 months post-transplantation. Everolimus (Certican) was administered orally, in two divided doses (b.i.d), and at the same time as Cyclosporine (Neoral). Everolimus (Certican) dose was adjusted in order to maintain a trough level between 3 and 8 ng/mL until randomization. Therefore, patients were randomized to cyclosporine withdrawal over a period of 1 month (±1 week) in study A2419 (NCT00154284) and over 3 months (±1 week) in study A2423 (NCT00170807). After randomization, final target trough range for everolimus was 8 - 12 ng/mL. Each patient was administered i.v. prednisone (or equivalent) pre- or intra-operatively according to center practice.
  Interventions: Drug: Everolimus (Certican); Drug: Cyclosporine (Neoral); Drug: Steroid; Drug: Basiliximab (Simulect)

INTERVENTIONS:
Drug: Everolimus (Certican)
  Other Names: Certican
Drug: Cyclosporine (Neoral)
  Other Names: Neoral
Drug: Steroid — Each patient was administered i.v. prednisone (or equivalent) pre- or intra-operatively according to center practice.
  Other Names: Prednisone
Drug: Basiliximab (Simulect)
  Other Names: Simulect

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of everolimus in combination with basiliximab, and steroids with and without cyclosporine microemulsion in de novo kidney transplant recipients.

DETAILED DESCRIPTION:
This is a combined analysis using 81 patients randomized and treated in CRAD001A2419 (NCT00154284) with 33 randomized and treated in CRAD001A2423 (NCT00170807). This approach is reflected in the protocol amendments for each study, and the one clinical study report for both.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of a first renal transplant from a primary cadaveric or non-HLA identical living related donor.
* Renal cold ischemic time < 36 hours.
* Age of donor < 65 years.

Exclusion Criteria:

* Patients who have received an investigational drug within 4 weeks of baseline period.
* Patients who are recipients of multiple organ transplants, including any organ other than kidney.
* Recipients of non-heart beating donor organs.

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2005-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis

REFERENCES:
- [Result] Grinyo JM, Paul J, Novoa P, et al. (2010). Better renal function in renal-transplant recipients treated with everolimus plus cyclosporine elimination compared with cyclosporine minimisation, Am J Transplant; 10(Suppl 4): 503: Abstract 1636.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from Spain from July 2005 to July 2008. As per protocol amendment, data were analyzed together with data from study CRAD001A2423 (NCT00154284) and CRAD001A2423 (NCT00170807).
Period: Overall Study
Arm/Group | Everolimus (Certican) With Cyclosporine (Neoral) Continuation | Everolimus (Certican) With Cyclosporine (Neoral) Withdrawal
Started | 59 ("Started" indicates Safety Population (randomized patients and treated after randomization.)) | 55
Intent to Treat (ITT) Population | 57 | 53
Completed | 52 ("Completed" means patients completed on study medication.All patients of both arms completed study.) | 42
Not Completed | 7 | 13
Not completed — Adverse Event | 6 | 9
Not completed — Abnormal laboratory value(s) | 0 | 1
Not completed — Lack of Efficacy | 1 | 2
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus (Certican) With Cyclosporine (Neoral) Continuation | Everolimus (Certican) With Cyclosporine (Neoral) Withdrawal | Total
Number analyzed (Participants) | 59 | 55 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (11.62) | 41.5 (12.27) | 43.6 (12.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 41 | 35 | 76

OUTCOME MEASURES:

1. Primary Outcome: Renal Function Measured by Calculated Glomerular Filtration Rate (GFR Calculated According to the Nankivell Formula)
Description: Nankivell's formula for calculated GFR is shown below:
  GFR [mL/min] = 6.7/C + W/4 - UREA/2 - 100/H2+ 35 (25 for females). Where W is body weight at specific visit [kg], H is height at specific visit [m], C is the serum concentration of creatinine [mmol/L], and UREA is the serum concentration of urea [mmol/L]. UREA was calculated from blood urea nitrogen (BUN) lab data by: UREA = 2.1441*BUN. If a GFR value from Nankivell formula was less than 10 [mL/min], then the value was assigned as 10 [mL/min].
Time Frame: At Month 3 and Month 12
Population: Intention to treat (ITT) population.
Measure: Mean (Standard Deviation); unit: mL/min per 1.73 m^2
Arm/Group | Everolimus (Certican) With Cyclosporine (Neoral) Continuation | Everolimus (Certican) With Cyclosporine (Neoral) Withdrawal
Number analyzed (Participants) | 57 | 53
mL/min per 1.73 m^2
  GFR at 3 months (Pre-randomization) | 68.5 (19.92) | 69.2 (18.40)
  GFR at 12 months | 63.6 (14.61) | 68.3 (15.13)

2. Secondary Outcome: Number of Participants With Biopsy-proven Acute Rejection (BPAR) Episodes, Graft Loss, Death or Loss to Follow-up
Description: Renal biopsies were collected for all cases of suspected acute rejection. For these cases, regardless of initiation of anti-rejection treatment, a graft core biopsy had been performed within 48 hours. These biopsies were listed on the Kidney Allograft Biopsy eCRF and the results used for patient management for BPAR. Graft loss was defined as the allograft was presumed to be lost on the day the patient started dialysis and was not able to subsequently be removed from dialysis as well as re-transplant. BPAR, graft loss, death, or loss to follow-up was analyzed by means of frequency tables.
Time Frame: Month 12
Population: Intention to treat (ITT) population.
Measure: Number; unit: Participants
Arm/Group | Everolimus (Certican) With Cyclosporine (Neoral) Continuation | Everolimus (Certican) With Cyclosporine (Neoral) Withdrawal
Number analyzed (Participants) | 57 | 53
Participants
  Biopsy-proven Acute Rejection (BPAR) | 10 | 10
  Graft Loss | 0 | 0
  Death | 0 | 0
  Loss to Follow-up | 0 | 0

3. Secondary Outcome: Serum Creatinine at Month 6 and 12
Description: serum creatinine summarized by mean and standard deviation
Time Frame: 6 month and 12 months
Population: Intention to treat (ITT) population.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Everolimus (Certican) With Cyclosporine (Neoral) Withdrawal | Everolimus (Certican) With Cyclosporine (Neoral) Continuation
Number analyzed (Participants) | 53 | 57
µmol/L
  6 Month | 120.1 (31.22) | 139.1 (47.03)
  12 Month | 123.0 (40.28) | 135.6 (40.61)

4. Secondary Outcome: Calculated Creatinine Clearance at 6 Month and 12 Month
Description: Creatinine clearance calculated by Cockcroft-Gault formula and summarized by mean, and standard deviation. Cockcroft-Gault formula to calculate Creatinine Clearance (CrCl[mL/min]) is shown below:
  CrCl[mL/min] = (140 - A) * W / (72 * C) * R. Where A is age at sample date [years], W is body weight at specific visit [kg], C is the serum concentration of creatinine [mg/dL], R = 1 if the patient is male and = 0.85 if female.
Time Frame: 6 month and 12 months
Population: Intention to treat (ITT) population.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Everolimus (Certican) With Cyclosporine (Neoral) Withdrawal | Everolimus (Certican) With Cyclosporine (Neoral) Continuation
Number analyzed (Participants) | 53 | 57
mL/min
  6 Month | 72.9 (19.34) | 63.6 (19.65)
  12 Month | 72.3 (20.50) | 65.6 (19.24)

ADVERSE EVENTS:
Arm/Group | Everolimus (Certican) With Cyclosporine (Neoral) Withdrawal | Everolimus (Certican) With Cyclosporine (Neoral) Continuation
Serious Adverse Events (participants affected / at risk) | 16/55 | 14/59
Other Adverse Events (participants affected / at risk) | 38/55 | 35/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (Certican) With Cyclosporine (Neoral) Withdrawal (N=55) | Everolimus (Certican) With Cyclosporine (Neoral) Continuation (N=59)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Transplant rejection (Immune system disorders) | 0 | 2
Abdominal wall infection (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Appendiceal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0
Febrile infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 2
Pneumonia (Infections and infestations) | 1 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Renal cyst infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 2
Soft tissue infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 3
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Renal lymphocele (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 3 | 0
Renal impairment (Renal and urinary disorders) | 0 | 2
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Lymphocele (Vascular disorders) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (Certican) With Cyclosporine (Neoral) Withdrawal (N=55) | Everolimus (Certican) With Cyclosporine (Neoral) Continuation (N=59)
Anaemia (Blood and lymphatic system disorders) | 5 | 8
Polycythaemia (Blood and lymphatic system disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 5
Oedema (General disorders) | 6 | 4
Oedema peripheral (General disorders) | 6 | 4
Pyrexia (General disorders) | 4 | 5
Bronchitis (Infections and infestations) | 1 | 3
Gastroenteritis (Infections and infestations) | 3 | 0
Nasopharyngitis (Infections and infestations) | 7 | 1
Urinary tract infection (Infections and infestations) | 5 | 9
Dyslipidaemia (Metabolism and nutrition disorders) | 4 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 6
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Proteinuria (Renal and urinary disorders) | 4 | 1
Renal impairment (Renal and urinary disorders) | 4 | 4
Acne (Skin and subcutaneous tissue disorders) | 4 | 0

LIMITATIONS AND CAVEATS:
This is a combined analysis using 81 patients randomized and treated in CRAD001A2419 with 33 randomized and treated in CRAD001A2423. This approach is reflected in the protocol amendments for each study, and the one clinical study report for both.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.